CLINICAL TRIAL: NCT03686020
Title: Sensitivity and Specificity of Serum and Salivary CYFRA21-1 in the Detection of Malignant Transformation in Oral Potentially Malignant Mucosal Lesions (Diagnostic Accuracy Study)
Acronym: CYFRA21-1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salsabeel Ali Mahmoud, PHD postgraduate student, Cairo University
Other Study IDs: 1152014
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Oral Potentially Malignant Lesions; Oral Cancer
Keywords: Oral potentially malignant lesions; Oral cancer; salivary CYFRA21-1; serum CYFRA21-1
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I: participants suffering from oral potentially malignant lesions
  Interventions: Diagnostic Test: Enzyme Linked Immunosorbent assay (ELISA)
- Group II: participants suffering from diagnosed oral malignant lesions
  Interventions: Diagnostic Test: Enzyme Linked Immunosorbent assay (ELISA)
- Group III: healthy participants who are systemically free, non-smokers, and not suffering from any oral mucosal lesions.
  Interventions: Diagnostic Test: Enzyme Linked Immunosorbent assay (ELISA)

INTERVENTIONS:
Diagnostic Test: Enzyme Linked Immunosorbent assay (ELISA) — measure serum and salivary CYFRA21-1 levels in all included participants using Enzyme Linked Immunosorbent assay (ELISA)

SUMMARY:
The study is designed to measure serum and salivary CYFRA21-1 levels using enzyme linked immunosorbent assay (ELISA) in patients with oral malignancy, oral potentially malignant lesions, and control subjects to evaluate the potential of CYFRA21-1 as a diagnostic marker for malignant transformation in potentially malignant oral mucosal lesions.

ELIGIBILITY:
Inclusion Criteria:

participants will be divided into 3 groups:

* Group I: patients suffering from oral potentially malignant lesions (PML) as defined by World Health Organization.
* Group II: patients suffering from diagnosed oral malignant lesions
* Group III: healthy subjects who are systemically free, non-smokers, and not suffering from any oral mucosal lesions.

Exclusion Criteria:

* Subjects taking any drugs inducing any changes that could affect the salivary flow.
* Pregnant females.
* Subjects have any allergies, infectious diseases or active dental abscesses during one month before saliva sampling.
* Patients receiving any drugs related to the oral lesions in the past 6 month prior to sample collection.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Egyptian population
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of serum and salivary CYFRA21-1 as a diagnostic marker in oral cancer | one year
  diagnostic accuracy in terms of sensitivity and specificity of serum and salivary CYFRA21-1 in differentiating between oral malignancy and oral potential malignant lesions in order to be able to early diagnose malignant changes in oral lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rajkumar K, Ramya R, Nandhini G, Rajashree P, Ramesh Kumar A, Nirmala Anandan S. Salivary and serum level of CYFRA 21-1 in oral precancer and oral squamous cell carcinoma. Oral Dis. 2015 Jan;21(1):90-6. doi: 10.1111/odi.12216. Epub 2013 Dec 30. PMID 24304502
- [Background] Alkotyfan K, Wiegand S, Muller HH, Windfuhr JP, Werner JA, Sesterhenn AM. Cyfra 21-1 as a tumor marker for follow-up of patients with squamous cell carcinoma of the oropharynx. Anticancer Res. 2010 Jun;30(6):2291-6. PMID 20651382
- [Background] Awasthi N. Role of salivary biomarkers in early detection of oral squamous cell carcinoma. Indian J Pathol Microbiol. 2017 Oct-Dec;60(4):464-468. doi: 10.4103/IJPM.IJPM_140_16. PMID 29323056
- [Background] Gualtero DF, Suarez Castillo A. Biomarkers in saliva for the detection of oral squamous cell carcinoma and their potential use for early diagnosis: a systematic review. Acta Odontol Scand. 2016;74(3):170-7. doi: 10.3109/00016357.2015.1110249. Epub 2015 Nov 18. PMID 26577643
- [Background] Malhotra R, Urs AB, Chakravarti A, Kumar S, Gupta VK, Mahajan B. Correlation of Cyfra 21-1 levels in saliva and serum with CK19 mRNA expression in oral squamous cell carcinoma. Tumour Biol. 2016 Jul;37(7):9263-71. doi: 10.1007/s13277-016-4809-4. Epub 2016 Jan 15. PMID 26779624
- [Background] Mortazavi H, Baharvand M, Mehdipour M. Oral potentially malignant disorders: an overview of more than 20 entities. J Dent Res Dent Clin Dent Prospects. 2014 Winter;8(1):6-14. doi: 10.5681/joddd.2014.002. Epub 2014 Mar 5. PMID 25024833
- [Background] Wang YX, Hu D, Yan X. Diagnostic accuracy of Cyfra 21-1 for head and neck squamous cell carcinoma: a meta-analysis. Eur Rev Med Pharmacol Sci. 2013 Sep;17(17):2383-9. PMID 24065233